CLINICAL TRIAL: NCT01252589
Title: Patient Reported Outcomes in Chronic Myeloid Leukemia. GIMEMA QoL - CML0310.
Brief Title: Patient Reported Outcomes in Chronic Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QoL - CML0310
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; Quality of Life; Symptoms; Patient-Reported outcomes; Questionnaire
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with CML: Adult patients (18 years of age or older) with confirmed diagnosis of CML
  Interventions: Other: HRQOL questionnaire

INTERVENTIONS:
Other: HRQOL questionnaire

SUMMARY:
Although the impact of disease and treatment related burden on health-related quality of life (HRQOL) in patients with solid tumours has been well studied, with several clinical trials that included HRQOL as an endpoint, the general understanding in patients with Chronic Myeloid Leukaemia (CML) is lacking in comparison.

The literature shows that patients' perspective is unique and should always be measured with methodologically sound instruments that are devised for this purpose.

The main scope of this project is develop to an international validated questionnaire for the purpose of HRQOL assessment; such a tool will then be used to provide important data, from the patients' perspective, to make more informed treatment decisions.

DETAILED DESCRIPTION:
The development process will follow the international guidelines published by the EORTC Quality of Life Group (QLG). This process will follow three main phases.

Phase 1 of will deal with the review of the literature, identification of an item list and interviews with experts in the treatment of CML and CML patients (undergoing all possible treatments).

In Phase II the identified issues from Phase I will be worded and translated into possible items for the provisional questionnaire using existing EORTC questionnaires and the EORTC QLG Item Bank.

In the Phase III the provisional CML questionnaire will be pre-tested by to a larger sample of CML patients (not the same patients involved in previous phases) and individual structured interviews will be conducted as well. These latter will identify questions that might be irrelevant or whether there will be additional issues not previously included.

Overall up to 480 patients will be enrolled in this study (up to 180 in phase I and up to 300 in phase III).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older)
* Confirmed diagnosis of Philadelphia chromosome positive CML
* Informed consent provided
* Patients enrolled in investigational treatment trials are eligible
* Ability to speak and read language of the Questionnaire

Exclusion Criteria:

* Freedom from overt cognitive impairment or major psychiatric conditions that may confound HRQOL evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years of age or older) with confirmed diagnosis of Philadelphia chromosome positive CML undergoing all possible treatments available.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2010-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Development of an EORTC questionnaire to assess HRQOL of patients with CML. | By the end of the study.

SECONDARY OUTCOMES:
Comparison between physicians' perception of relevance of HRQOL issues with that of patients. | By the end of the study.
Development of an EORTC CML symptom checklist. | By the end of the study.
HRQOL in CML patients undergoing 2nd line treatment with TKIs. | By the end of the study.
Decision making process for choosing between different 2nd line treatments with TKIs. | By the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, PhD, Principal Investigator — GIMEMA DATA CENTER, ROME, ITALY
Locations (14):
- Dana-Farber Cancer Institute Harvard University, Boston, Massachusetts, United States
- Innsbruck University Hospital, Innsbruck, Austria
- University of Ghent, Ghent, Belgium
- Centre Hospitalier Universitaire of Poitiers, Poitiers, France
- University of Heidelberg, Heidelberg, Germany
- University of Athens, Athens, Greece
- University of Baghdad, Baghdad, Iraq
- Italy (5):
  - Policlinico S. Orsola - Malpighi, Università di Bologna, Bologna
  - Ematologia Ospedale "Binaghi", Cagliari, Cagliari
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Ospedale S.Maria delle Croci, Ravenna
  - Ematologia - Sapienza Università di Roma, Roma
- Tilburg University, Tilburg, Netherlands
- National Taiwan University, Taipei, Taiwan

REFERENCES:
- [Background] Efficace F, Baccarani M, Breccia M, Saussele S, Abel G, Caocci G, Guilhot F, Cocks K, Naeem A, Sprangers M, Oerlemans S, Chie W, Castagnetti F, Bombaci F, Sharf G, Cardoni A, Noens L, Pallua S, Salvucci M, Nicolatou-Galitis O, Rosti G, Mandelli F. International development of an EORTC questionnaire for assessing health-related quality of life in chronic myeloid leukemia patients: the EORTC QLQ-CML24. Qual Life Res. 2014 Apr;23(3):825-36. doi: 10.1007/s11136-013-0523-5. Epub 2013 Sep 13. PMID 24026634
- See also: GIMEMA — http://www.gimema.it